CLINICAL TRIAL: NCT05249192
Title: Immediate Versus Early (24-hours) Urinary Catheter Removal After Elective Minimally Invasive Colonic Resection: Study Protocol for a Randomized, Multicenter, Non-inferiority Trial
Brief Title: Immediate Versus Early (24-hours) Urinary Catheter Removal After Elective Minimally Invasive Colonic Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Faenza Hospital (Unknown); Ravenna Hospital (Unknown); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other); Humanitas University (Other); Universita di Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EURiCaRe
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Surgical Complication; Colonic Disease; Postoperative Complications; Urinary Retention Postoperative; Urinary Tract Infections
MeSH Terms: conditions — Colonic Diseases; Postoperative Complications; Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled, two-arm, multi-center trial
Who Masked: Participant, Care Provider
Masking Description: patients and surgeons are blinded to group allocation until the end of surgical procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate UC removal (Experimental): Urinary catheter removal immediately after the end of the surgical procedure before exiting the operating room.
  Interventions: Device: Immediate urinary catheter removal
- Early UC removal (Active Comparator): Urinary catheter removal on first postoperative day (6 a.m.) as per standard protocol
  Interventions: Device: Early urinary catheter removal

INTERVENTIONS:
Device: Immediate urinary catheter removal — Urinary catheter removal immediately after the end of the surgical procedure before exiting the operating room.
  Arms: Immediate UC removal
Device: Early urinary catheter removal — urinary catheter removal on the first postoperative day (6 a.m)
  Arms: Early UC removal

SUMMARY:
The primary aim of this study is to compare the rate of acute urinary retention (AUR) after immediate compared to early (24-hours) removal of urinary catheter (UC) in patients undergoing minimally invasive colorectal resection. The study hypothesis is that immediate UC removal is non-inferior to 24-hours UC removal in terms of AUR rate.

The secondary outcomes focus on goals that could be positively impacted by the immediate removal of the UC at the end of the surgery. In particular, the rate of urinary tract infections, perception of pain, time-to-return of bowel and physical functions, postoperative complications and postoperative length of stay will all be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 years and 80 years old
2. Patients scheduled to undergo minimally invasive resection of the colon under general anesthesia
3. Willingness to participate
4. Compliance to study purpose
5. Written informed consent

Exclusion Criteria:

1. Need for an anastomosis below the anterior peritoneal reflection
2. Need for a major resection other than colorectal
3. Need for post-operative intensive care monitoring or intensive care unit (ICU) stay
4. Anesthesia time longer than 300 minutes
5. Presence of chronic indwelling UC
6. Presence of an entero-vesical fistula
7. Need for ureteral stent placement, bladder resection or repair
8. A previous and unsolved history of AUR or overt voiding dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Acute urinary retention rate | 3 days postoperatively
  Occurrence of urinary retention after removal of urinary catheter

SECONDARY OUTCOMES:
Urinary tract infections | 30 days postoperatively
  Occurrence of urinary tract infections
UC reinsertion | 30 days postoperatively
  need for urinary catheter reinsertion after first removal
Pain scores | 6,12,24,48 and 72 hours after surgery
  Numeric Rating Scores (NRS) for abdominal pain (0-10)
Bowel function | 10 days postoperatively
  Time for return of bowel function as for flatus and stools postoperatively
Mobilization | 10 days postoperatively
  Return to passive and active mobilization postoperatively
Morbility | first 30 days after surgery
  Postoperative morbility according to the Clavien-Dindo classification
Length of hospital stay | 30 days postoperatively
  postoperative stay

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Pedrazzani, Professor, Principal Investigator — Universita di Verona
Locations (1):
- Division of General and Hepatobiliary Surgery, Verona, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedrazzani C, Montroni I, Conti C, Turri G, Foppa C, Carvello M, Taffurelli G, Ugolini G, Spinelli A. Immediate versus early (24-hours) urinary catheter removal after elective minimally invasive colonic resection: study protocol for a randomized, multicenter, non-inferiority trial. Trials. 2022 Nov 22;23(1):956. doi: 10.1186/s13063-022-06894-6. PMID 36414969